CLINICAL TRIAL: NCT00584259
Title: Effect of Coffee on Gastro-Esophageal Disease in Patients With Symptoms of Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Peter Belafsky, MD, Ph.D., University of California Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 200614348-2
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: GERD
Keywords: GERD; Gastro-Esophageal Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Coffee — 3 cups of coffee over a 24 hour period

SUMMARY:
Investigation evaluating the effect of coffee on gastro-esophageal reflux disease.

DETAILED DESCRIPTION:
Many patients with gastro-esophageal reflux disease (GERD) report that drinking coffee causes heartburn. The purpose of this study is to investigate the effects of coffee on gastro-esophageal acid reflux, and its relation to esophageal motility parameters in patients who are already scheduled to undergo 48 hour wireless pH testing as a result of having symptoms suggestive of GERD. The specific aims are to evaluate the effects of coffee on GERD during daily life and to elucidate the underlying pathogenic mechanism by which coffee induces reflux.

ELIGIBILITY:
Inclusion Criteria:

* persons undergoing wireless pH testing for diagnosis and treatment of GERD

Exclusion Criteria:

* those under the age of 18
* pregnant and lactating women
* those who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
coffee leads to reflux events | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States